CLINICAL TRIAL: NCT05555940
Title: Study on the Effect and Brain Influence Mechanism of Individualized Precise Transcranial Magnetic Stimulation Based on Image Analysis on Emotional Blunting in Depression
Brief Title: Effect of Individualized Precise TMS on Emotional Blunting in Depression and Its Brain Imaging Mechanism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XJLL-KY20222175
Record Dates: First submitted 2022-09-13; First posted 2022-09-27 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2023-12

CONDITIONS: Depression
Keywords: emotional blunting; transcranial magnetic stimulation
MeSH Terms: conditions — Depression | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TMS true stimulation group (Experimental): Transcranial magnetic stimulation and medication. The stimulation parameters were 10Hz frequency and 120%MT intensity. 50 treatment sequences were given each time, with 60 stimulation times for each sequence, the sequence interval was 30 seconds, and a total of 3000 stimulation times for each treatment. The patients were treated once a day for 15 days. Medical treatment is selective serotonin reuptake inhibitors/serotonin-noradrenaline reuptake inhibitors (SSRIs/SNRIs).
  Interventions: Device: Transcranial magnetic stimulation
- TMS sham stimulation group (Sham Comparator): Sham stimulation and medication. The pseudo-stimulation method was to flip the magnetic head at 90 degrees with the scalp, The stimulation parameters were 10Hz frequency and 120%MT intensity. 50 treatment sequences were given each time, with 60 stimulation times for each sequence, the sequence interval was 30 seconds, and a total of 3000 stimulation times for each treatment. The patients were treated once a day for 15 days. Medical treatment is selective serotonin reuptake inhibitors/serotonin-noradrenaline reuptake inhibitors (SSRIs/SNRIs).
  Interventions: Device: Transcranial magnetic stimulation

INTERVENTIONS:
Device: Transcranial magnetic stimulation — The stimulation sites of the true TMS group were mPFC-amygdala functional junction and SSRIs/SNRIs treatment, while the sham TMS group was treated with reversed magnetic head sham stimulation and SSRIs/SNRIs treatment.
  Other Names: SSRIs/SNRIs

SUMMARY:
This study aims to explore and investigate the therapeutic effect and mechanism of individualized localization of transcranial magnetic stimulation on emotional blunting of depression, improve the understanding of the mechanism of emotional blunting of depression, order to provide new treatment methods and better curative effects for this disease.

DETAILED DESCRIPTION:
Depression is a common mental illness. The traditional treatment is medication, but many patients do not respond well to medication and have side effects such as emotional blunting. emotional blunting is a numbness to both positive and negative emotions. It is estimated that about 40% to 60% of depressed patients who use serotonin (5-HT) reuptake inhibitors (SSRIs) or 5-HT and norepinephrine (NE) reuptake inhibitors (SNRIs) have varying degrees of affective retardation. Repetitive transcranial magnetic stimulation (rTMS) is a safe and non-invasive method for the treatment of depression. Its clinical efficacy is related to the accuracy of the stimulation target. How to carry out individualized accurate positioning is of great significance for improving the therapeutic effect.

ELIGIBILITY:
Inclusion Criteria:

* (1) Outpatients of all genders, aged ≥18 years and ≤65 years, right-handed, admitted to the psychosomatic Department of Xijing Hospital;

  (2) In accordance with the diagnostic criteria for the depressive disorder of the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V)).

  (3) Montgomery-Asberg Depression Rating Scale (MADRS): total MADRS score ≥12;

  (4) The total score of the Oxford Depression Questionnaire (ODQ) at baseline was ≥50, and the answer to the standardized screening question of emotional blunting was "yes";

  (5) Received at least 6 weeks of monotherapy with an SSRI or SNRI prior to enrollment;

  (6) Subjects who can understand and are willing to strictly follow the clinical trial protocol to complete this study and sign informed consent.

Exclusion Criteria:

* (1) Have a history of substance abuse within 6 months before the start of the study;

  (2) Patients with bipolar disorder and depression caused by other mental diseases (such as psychoactive substances and non-dependent substances);

  (3) Have a history of somatic severe diseases or diseases that may affect the central nervous system (such as tumors, syphilis, etc.);

  (4) Have neurological diseases or risk of seizures, such as previous brain diseases, head trauma, alcoholism, EEG abnormalities, MRI evidence of abnormal brain structure, or family history of epilepsy;

  (5) There are contraindications to MRI scanning or transcranial magnetic stimulation treatment, such as metal or electronic instruments (intracranial metal foreign bodies, cochlear implants, cardiac pacemakers, stents, and other metal foreign bodies);

  (6) Have obvious suicide risk, or have actual suicide behavior within 6 months before the start of the study;

  (7) Pregnant, breastfeeding, or planning pregnancy during the trial;

  (8) Other conditions that are not suitable for the study object in the researcher's judgment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes from Baseline on Oxford Depression Questionnaire scores during treatment and at each follow-up point. | At baseline, at the end of treatment on day 7, at the end of treatment on day 15, 2 weeks after treatment, 4 weeks after treatment, and 8 weeks after treatment
  The Oxford Depression Questionnaire(ODQ) is a relatively new tool for assessing emotional retardation, a self-rating scale.It includes three sections and 26 questions, focusing on the emotional experience of patients in the past week.Each question is scored on a 5-point scale from 1 (disagree) to 5 (agree). And summarized into a score for each dimension and a total score (total score range: 26-130). The higher the value on ODQ, the higher the level of emotional blunting.

SECONDARY OUTCOMES:
Changes from Baseline on Montgomery-Asberg Depression Rating Scale scores or other clinical scales during treatment and at each follow-up point. | At baseline,at the end of treatment on day 7, at the end of treatment on day 15, 2 weeks after treatment, 4 weeks after treatment, and 8 weeks after treatment
  There are 10 items in the Montgomery-Asberg Depression Rating Scale（MADRS）, and each item is divided into 6 levels according to the identity level, with a score of 0-6 points. The total score of patients is 0-60. The higher the score of patients, the more severe the depression.
Changes of MRI from baseline to the end of 15 day treatment period. | Before treatment, 15 days
  Before and after treatment, MRI is performed for each patient to measure the blood oxygen level of each brain region, from which the functional connectivity between brain regions could be statistically obtained, and then the differences of the functional connectivity before and treatment are compared.

CONTACTS AND LOCATIONS:
Locations (1):
- XijingH, Xi'an, Shannxi, China

REFERENCES:
- [Derived] Zhang Y, Tang N, Lei L, Lv R, Zhang Y, Liu N, Chen H, Cai M, Wang H. Efficacy of functional magnetic resonance imaging-guided personalized repetitive transcranial magnetic stimulation (fMRI-rTMS) in depressive patients with emotional blunting: study protocol for a randomized controlled trial. Trials. 2024 Feb 21;25(1):134. doi: 10.1186/s13063-024-07976-3. PMID 38383418